CLINICAL TRIAL: NCT04528420
Title: Evaluation of Optimised Early Management in the Context of Radiochemotherapy for Curatively Treated Squamous Cell Carcinoma of the Head and Neck
Brief Title: Optimised Early Management of Squamous Cell Carcinoma of the Head and Neck Cancer
Acronym: OPTINECK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHB19.01
Record Dates: First submitted 2020-07-29; First posted 2020-08-27 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
Keywords: radiochemotherapy; nutrition; support care; early management
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimised arm (Experimental): Patients will be taken care of early and optimally way.
  Interventions: Other: optimised management
- Standard arm (No Intervention): Patients will be monitored as in standard practice

INTERVENTIONS:
Other: optimised management — At the inclusion , the patient will benefit from an early consultation with a nutritionist, a pain doctor and a social worker.
  During the preparation phase for radiotherapy the patient will benefit from weekly consultations with a pain nurse and a dietician.
  During the radiotherapy the patient will be weighed daily and have an assessment of their nutritional needs and a weekly consultation with a pain nurse and dietician and then twice a month until three months post-radiotherapy.
  Arms: Optimised arm

SUMMARY:
Post-operative concomitant radiochemotherapy is a treatment that is difficult to achieve for several reasons. First of all, and by definition, these patients have had recent surgery, most often accompanied by several weeks of hospitalization and weight loss. In addition, the functional recovery of feeding capacity is not always complete at the time of the start of irradiation. In addition, concomitant radiochemotherapy is responsible for very frequent radiomucitus which alters the feeding capacity of patients during treatment.

In total, the rate of complete radiochemotherapy (3 cures of cisplatin administered) varies from 50 to 70% depending on the studies, which were carried out in selected populations within the framework of an experimental clinical trial and without distinguishing between positive and negative Human Papilloma tumours . In our experience, in a population with a very high preponderance of non-Human Papilloma-related tumours and not selected by participation in an experimental trial, complete radiochemotherapy is only possible in about 40% to 50% of cases.However, the amount of cisplatin actually administered is correlated with overall survival. Therefore, it is logical to assume that increasing the number of patients receiving full treatment may result in increased survival.

While the need for nutritional care during radiotherapy is clearly established, its modality remains debated. Recently, a randomised study of 159 patients treated by radiotherapy (or radiochemotherapy) showed that the simple systematic prescription of oral food supplements (500 kcal/d) in addition to the usual dietary advice was associated with a lesser reduction in weight at the end of radiotherapy (main objective) but also with an improvement in the tolerance of the treatments. Overall, nutritional management during treatment varies greatly, ranging from simple dietary monitoring to prophylactic gastrostomy and the insertion of a nasogastric tube on demand during treatment. This heterogeneity of management found in the literature is also observed at the regional level. This project will also make it possible to propose a harmonized support strategy at the inter-regional level.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, over 18 and under 75 years of age,
* Worl Health Organisation score < 2,
* Treatment for a localized squamous cell carcinoma of the head and neck for which a curative treatment by concomitant post-operative radiochemotherapy based on cisplatin is retained,
* Having signed the informed consent,
* Affiliate or beneficiary of a social protection scheme.

Exclusion Criteria:

* History of other neoplastic disease less than 2 years old or progressive,
* History of radiotherapy for head and neck cancer,
* Contraindications to cisplatin,
* Pregnant or breastfeeding woman,
* Protected major (under guardianship or curatorship),
* Patient participating in a therapeutic study
* Patient unable to understand the study for any reason or to comply with the constraints of the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2020-11-26 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Assessing of the impact of early multimodal management on weight loss measured between the inclusion consultation and 3 months post-treatment. | 3 months post treatment
  Proportion of patients with at least 5% reduction in weight at 3 months post-treatment compared to the inclusion consultation

SECONDARY OUTCOMES:
Assessing the impact of multimodal management on overall survival and progression-free survival at 18 months post-treatment | 18 months post treatment
  Overall and progression-free survival rate at 18 months post-treatment
Assessing the impact of multimodal management on the percentage of patients receiving the full treatment as planned | 1 month
  Percentage of patients who received all the treatment as planned
Assessing the impact of multimodal management on the percentage of patients receiving level 3 analgesics during radio-chemotherapy and up to 3 months post-treatment | 3 months post treatment
  Number of patients who level 3 analgesics has been prescribed
Assessing the impact of multimodal management on average weight loss | 18 months post treatment
  Average of difference of weight at the end of the study and weight at the inclusion
Medico-economic analysis of multimodal management using the cost-utility method | 18 months post treatment
  Cost-utility ratio in each arm

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Thureau, MD,PhD, Study Director — Centre Henri Becquerel
Locations (7):
- France (7):
  - CHU Amiens, Amiens
  - CH Beauvais, Beauvais
  - Clinique du Parc, Caen
  - Centre Guillaume le Conquérant, Le Havre
  - CHRU Lille, Lille
  - Centre Henri Becquerel, Rouen
  - CH Saint-Quentin, Saint-Quentin

IPD SHARING:
Plan to Share IPD: No